CLINICAL TRIAL: NCT04128813
Title: A Comparison of the Effect of Two Types of Whole Body Vibration on Fibromyalgia. A Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IB 2586/15 PI-2
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: In this clinical trial design, three groups of participants receive different interventions. One group receives a training with a vertical whole body vibration plattform, another group receives a training with a rotational whole body vibration platform and the third one is the control group.
Who Masked: Participant, Investigator
Masking Description: In this clinical trial design strategy, the participants and the investigator do not know which participants have been assigned which interventions so there is a double-blind masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vertical whole body vibration platform. (Active Comparator): Use of a rotational whole body vibration platform.
  Interventions: Device: Vertical whole body vibration
- Rotational whole body vibration platform (Active Comparator): Use of a rotational whole body vibration platform.
  Interventions: Device: Vertical whole body vibration
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Device: Vertical whole body vibration — A neuromuscular treatment using two types of whole body vibration platforms, a rotational and a vertical platform.
  Other Names: Rotational whole body vibration
  Arms: Rotational whole body vibration platform; Vertical whole body vibration platform.

SUMMARY:
The objective of this study is to compare the effectiveness of two types of body vibration platform, one vertical and one rotational, through a 12-week training in patients with fibromyalgia.

DETAILED DESCRIPTION:
This is a single blind randomized controlled trial. Sixty patients of FM will be assigned randomly to 3 study groups: 20 patients will be part of the vertical whole body vibration experimental group in the EG1, that will perform a neuromuscular treatment using the vertical whole body vibration platform, another 20 will constitute the rotational whole body vibration experimental group in the EG2, that will perform a neuromuscular treatment using the rotational whole body vibration platform, and another 20 will constitute the control group (CG). All these subjects will sign the corresponding informed consent for their participation in the study, according to the ethical criteria established in the Helsinki Declaration. The study will take place between January and December 2016. Three groups of variables were analyzed in the present study three times: before, after and follow-up after three months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of fibromyalgia according with the 1990 classification criteria of the American College of Rheumatology for fibromyalgia

Exclusion Criteria:

* History of severe trauma.
* Severe disease that prevents supporting the program physical load.
* Pregnancy.
* Participation in a psychological or physical therapy program.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-01-17 (Estimated); Study Completion 2020-04-17 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Thresholds | 20 minutes
  Pressure stimuli were applied on epicondyles and index finger.
Vibration Thresholds | 20 minutes
  Peripheral sensory function was evaluated by measuring vibration thresholds.
Six-minute Walking Test (6MWT) | 6 minutes.
  The 6MWT is a functional test in which the patient walks what he can during 6 minutes, analyzing the total distance walked.
Dynamometer | 5 minutes.
  A back muscle dynamometer was used to measure isometric back muscle strength.
Romberg's Balance Test Modified Version | 1 minute.
  In the present study, we analyzed the oscillatory body movements during the test performance. Participants were situated below a cam situated above the ground and regulated to be placed at a mean distance of 50 cm. from the participant's head. They were asked to remain in orthostatic position with feet parallel at shoulder height, arms extended along the body and eyes closed for 1 minute.
Gait Task | 5 minutes.
  gait velocity (cm/sec)
Fibromyalgia Impact Questionnaire (FIQ) | 10 minutes.
  Fibromyalgia Impact Questionnaire (FIQ
Visual Analogue Pain Scale (VAS) | 5 minutes.
  Each participant was asked to indicate their current level of pain using a 20 cm VAS that ranged from 0 (no pain) to 100 (highest level of pain).
Perceived Quality of Life Index | 10 minutes.
  The Quality of Life Index (QLI-Sp) is a self-report questionnaire that measures perceived health-related quality of life that includes 10 items or domains: physical wellbeing, psychological/emotional well-being, selfcare and independent functioning, occupational functioning,interpersonal functioning, social-emotional support, community and services support, personal fulﬁlment, spiritual fulﬁlment, and overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio JA Mingorance, PhD, Study Chair — Professor
Locations (1):
- University of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanudo B, de Hoyo M, Carrasco L, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, McVeigh JG. Effect of whole-body vibration exercise on balance in women with fibromyalgia syndrome: a randomized controlled trial. J Altern Complement Med. 2012 Feb;18(2):158-64. doi: 10.1089/acm.2010.0881. Epub 2012 Feb 9. PMID 22321155
- [Result] Adsuar JC, Del Pozo-Cruz B, Parraca JA, Olivares PR, Gusi N. Whole body vibration improves the single-leg stance static balance in women with fibromyalgia: a randomized controlled trial. J Sports Med Phys Fitness. 2012 Feb;52(1):85-91. PMID 22327091